CLINICAL TRIAL: NCT05943860
Title: Efficacy and Tolerability of Pantovigar® Vegan in Female Subjects With Diffuse Hair Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz Pharmaceuticals GmbH (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M900411001
Record Dates: First submitted 2023-06-21; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Diffuse Hair Loss in Females

STUDY DESIGN:
Intervention Model Description: Intra-individual comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pantovigar vegan treatment (Experimental)
  Interventions: Dietary Supplement: Pantovigar® vegan

INTERVENTIONS:
Dietary Supplement: Pantovigar® vegan — Oral application of 1 capsule three times a day (morning, noon, evening) for 6 months

SUMMARY:
The objective of this study is to assess the hair growth efficacy of a Food for Special Medicinal Purposes (FSMP) Pantovigar® vegan after 3 and 6 months of intake.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse hair loss
* Modified Savin Score I to III
* Hair length of at least 2 cm

Exclusion Criteria:

* Pathological hair loss (like alopecia areata, universalis or totalis; scarring alopecias; androgenic alopecia; inflammatory conditions of the scalp)
* Symptomatic diffuse alopecia due to pathological low iron concentration or thyroid gland disorder
* Acute telogen effluvium
* Recent or concomitant treatment with any drugs that may cause hair loss
* Concomitant diseases that can cause hair loss

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Self-assessment questionnaire for product acceptance by subjects | Months 3
Self-assessment questionnaire for product acceptance by subjects | Months 6

SECONDARY OUTCOMES:
Effect on hair growth assessed by phototrichogram analysis | Baseline up to month 6
Change from baseline of blood parameters: Ferritin | Baseline up to month 6
Change from baseline of several blood parameters: Vitamin B1 | Baseline up to month 6
Change from baseline of several blood parameters: Biotin | Baseline up to month 6
Change from baseline of several blood parameters: Folic acid | Baseline up to month 6
Change from baseline of several blood parameters: Hematocrit | Baseline up to month 6
Change from baseline of several blood parameters: Pantothenic Acid | Baseline up to months 6
Occurrence of treatment-emergent adverse reactions and treatment-emergent serious adverse reactions | Baseline up to months 6

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Therapeutics
Locations (1):
- proDerm, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No